CLINICAL TRIAL: NCT07402720
Title: Clinical Effectiveness Of Polishing Brush Compared to Ceramic Soft Tissue Trimming Bur In Gingival Depigmentation: A Randomized Controlled Trial
Brief Title: Clinical Effectiveness Of Polishing Brush Compared To Ceramic Soft Tissue Trimming Bur In Gingival Depigmentation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Raghad hisham, Principal Investigator Raghad Hisham, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2026PER3-3-1
Record Dates: First submitted 2026-01-25; First posted 2026-02-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gingival Hyperpigmentation
Keywords: ceramic bur; polishing brush; gingival hyperpigmentation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polishing brush (Active Comparator): In the test group, gingival depigmentation will be performed using a polishing brush specifically adapted for soft tissue application. After administering local anesthesia, a silicon carbide or rubber-based polishing brush will be attached to a low-speed handpiece. The pigmented gingival epithelium will be gently abraded in a circular motion under light pressure until the superficial pigmented layer is removed and uniform pink gingiva is visible. Continuous irrigation with sterile saline will be used to prevent heat generation and ensure visibility. The operator will take care not to injure the underlying connective tissue. No periodontal dressing will be applied. Postoperative instructions will include gentle oral hygiene, avoiding hot or spicy foods, and use of 0.12% chlorhexidine mouthwash for 1 week.
  Interventions: Procedure: Gingival Depigmentation using polishing brush
- Ceramic bur (Experimental): In the control group, ceramic soft tissue trimming burs will be used to perform gingival depigmentation. After achieving local anesthesia, a flame- or round-shaped ceramic bur will be attached to a low-speed contra-angle handpiece. The bur will be used in a brushing motion to carefully remove the pigmented epithelial layer without applying excessive pressure. The clinician will maintain light, controlled strokes to avoid damaging the underlying lamina propria. As with the polishing brush technique, continuous irrigation with saline will be provided to cool the tissue and improve visibility. Once the pigmented areas are cleared and a healthy pink gingival color is achieved, the procedure will be concluded without any periodontal dressing. Postoperative care will follow the same protocol as the polishing brush group.
  Interventions: Procedure: Depigmentation using ceramic soft tissue trimming bur

INTERVENTIONS:
Procedure: Gingival Depigmentation using polishing brush — gingival depigmentation will be performed using a polishing brush specifically adapted for soft tissue application. After administering local anesthesia, a silicon carbide or rubber-based polishing brush will be attached to a low-speed handpiece. The pigmented gingival epithelium will be gently abraded in a circular motion under light pressure until the superficial pigmented layer is removed and uniform pink gingiva is visible. Continuous irrigation with sterile saline will be used to prevent heat generation and ensure visibility. The operator will take care not to injure the underlying connective tissue. No periodontal dressing will be applied. Postoperative instructions will include gentle oral hygiene, avoiding hot or spicy foods, and use of 0.12% chlorhexidine mouthwash for 1 week.
  Arms: Polishing brush
Procedure: Depigmentation using ceramic soft tissue trimming bur — ceramic soft tissue trimming burs will be used to perform gingival depigmentation. After achieving local anesthesia, a flame- or round-shaped ceramic bur will be attached to a low-speed contra-angle handpiece. The bur will be used in a brushing motion to carefully remove the pigmented epithelial layer without applying excessive pressure. The clinician will maintain light, controlled strokes to avoid damaging the underlying lamina propria. As with the polishing brush technique, continuous irrigation with saline will be provided to cool the tissue and improve visibility. Once the pigmented areas are cleared and a healthy pink gingival color is achieved, the procedure will be concluded without any periodontal dressing. Postoperative care will follow the same protocol as the polishing brush group.
  Arms: Ceramic bur

SUMMARY:
Gingival hyperpigmentation, particularly of melanin origin, can pose significant aesthetic concerns, especially among patients with a high smile line. Several depigmentation techniques have been proposed to manage this condition, including scalpel surgery, electrosurgery, cryotherapy, lasers, and various rotary instruments. Recently, minimally invasive rotary tools such as ceramic burs and polishing brushes have gained interest due to their potential to deliver controlled ablation with reduced postoperative discomfort and healing complications.

Ceramic soft tissue trimming burs are specially designed to remove superficial pigmented gingival layers with minimal trauma. However, these instruments may still generate heat and cause a degree of tissue damage. On the other hand, polishing brushes, traditionally used for surface finishing and stain removal, have recently been explored for soft tissue applications due to their gentle action and adaptability.

Despite their increasing use, there is insufficient comparative clinical evidence on the efficacy, healing outcomes, and patient-centered experiences between these two modalities in gingival depigmentation. A split-mouth randomized controlled trial design offers the advantage of eliminating inter-individual variability. Thus, this study aims to assess and compare the clinical effectiveness of the polishing brush and ceramic trimming bur for gingival depigmentation in terms of pigment reduction, healing outcomes, postoperative pain, and recurrence.

DETAILED DESCRIPTION:
This study is designed as a prospective randomized controlled clinical trial with a parallel intraoral comparison between two treatment modalities:

1. Depigmentation using polishing brush and
2. Depigmentation using ceramic soft tissue trimming bur. Participants will be randomly allocated into two independent groups, with each group receiving one of the two interventions on both sides of the arch. This parallel design ensures that each participant receives only one treatment modality, thereby preventing any crossover effects and allowing for between-subject comparison. Randomization will be conducted using a computergenerated sequence to ensure unbiased allocation. Blinding of the outcome assessor will be maintained to minimize assessment bias.

The trial will adhere to CONSORT guidelines, with baseline data collection followed by standardized clinical evaluations at predefined follow-up intervals to assess changes in gingival thickness and other relevant soft tissue parameters.

The study will be conducted at the Department of Oral Medicine and Periodontology, Faculty of Dentistry - Cairo University, Egypt.

Participants will be recruited from the outpatient clinic of the same department.

Population:

Systemically healthy patients with gingival hyperpigmentation.

Intervention:

Depigmentation using a polishing brush.

Comparison:

Depigmentation using ceramic soft tissue trimming bur.

Treatment:

Healthy, nonsmokers with moderate to severe gingival hyperpigmentation in both arches will be assigned for Polishing Brush Compared To Ceramic Soft Tissue Trimming Bur • Study Groups:

* Group 1: Depigmentation using polishing brush
* Group 2: Depigmentation using ceramic soft tissue trimming bur

Preoperative evaluation:

1. Clinical examination: A comprehensive clinical examination of the patient's oral cavity and periodontal condition will be performed to assess baseline oral health. This will be complemented by a structured oral interview aimed at evaluating the patient's adherence to the study's inclusion criteria, with a particular focus on oral hygiene practices, habits and overall compliance.

Polishing brush In the test group, gingival depigmentation will be performed using a polishing brush specifically adapted for soft tissue application.

After administering local anesthesia, a silicon carbide or rubber-based polishing brush will be attached to a low-speed handpiece. The pigmented gingival epithelium will be gently abraded in a circular motion under light pressure until the superficial pigmented layer is removed and uniform pink gingiva is visible. Continuous irrigation with sterile saline will be used to prevent heat generation and ensure visibility. The operator will take care not to injure the underlying connective tissue. No periodontal dressing will be applied. Postoperative instructions will include gentle oral hygiene, avoiding hot or spicy foods, and use of 0.12% chlorhexidine mouthwash for 1 week.

Ceramic bur In the control group, ceramic soft tissue trimming burs will be used to perform gingival depigmentation. After achieving local anesthesia, a flame- or round-shaped ceramic bur will be attached to a low-speed contra-angle handpiece. The bur will be used in a brushing motion to carefully remove the pigmented epithelial layer without applying excessive pressure. The clinician will maintain light, controlled strokes to avoid damaging the underlying lamina propria. As with the polishing brush technique, continuous irrigation with saline will be provided to cool the tissue and improve visibility. Once the pigmented areas are cleared and a healthy pink gingival color is achieved, the procedure will be concluded without any periodontal dressing. Postoperative care will follow the same protocol as the polishing brush group.

Patient-Reported Outcomes:

Oral health-related quality of life (OHRQoL) will be assessed using the validated Oral Health Impact Profile (OHIP-14) questionnaire, which measures the functional, psychological, and social impacts of oral conditions on everyday life. The OHIP-14 consists of 14 items covering seven conceptual domains: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. Participants will complete the OHIP-14 at baseline and again three months post-treatment to assess changes in self-perceived oral health status and quality of life. Incorporating this patient-reported outcome measure enables a comprehensive evaluation of treatment effectiveness beyond clinical indicators alone.

Postoperative instructions and follow up:

All patients will receive standardized postoperative care instructions immediately following the depigmentation procedure. Patients will be advised to avoid trauma or mechanical irritation to the treated area for at least 1-2 weeks. Toothbrushing in the surgical sites will be restricted to the use of an ultrasoft toothbrush, and gentle brushing techniques will be demonstrated. The use of chemical plaque control agents such as 0.12% chlorhexidine mouthwash will be prescribed twice daily for 1-2 weeks to aid plaque control and reduce the risk of postoperative infection.

Patients will be instructed to refrain from consuming hot, spicy, or abrasive foods for the first few days to minimize discomfort and irritation. Analgesics will be prescribed as needed for pain management, according to individual patient tolerance and medical history.

Postoperative Follow-Up :

Patients will be recalled for clinical evaluation at 1 week, 2 weeks, 1 month, and 3 months postoperatively. At each follow-up visit, the surgical sites will be examined for signs of healing, presence of infection, inflammation, or any adverse tissue reactions. Re-epithelialization, color match with surrounding gingiva, patient comfort, and recurrence of pigmentation will be assessed and documented.

Professional plaque control will be reinforced at each visit, and oral hygiene instructions will be reiterated as necessary. Any complications or patient-reported concerns will be addressed promptly.

If re-pigmentation is noted during the follow-up period, its extent and pattern will be recorded for further analysis. Digital photographs may be taken at baseline and each follow-up visit to monitor healing and pigmentation changes objectively.

ELIGIBILITY:
Inclusion Criteria:

* Presence of melanin hyperpigmentation (Dummett Oral Pigmentation Index ≥ 2)
* Presence of bilateral gingival pigmentation extending at least 3 teeth in each arch
* Age range: e.g., 18-40 years (adjust based on your sample)
* Non-smokers (or smokers <10 cigarettes/day, specify if allowed)
* Systemically healthy
* Willingness to participate and sign informed consent 8
* Available for follow-up appointments
* No previous periodontal surgery in the area other than prophylaxis

Exclusion Criteria:

* • Systemic conditions affecting healing (e.g., diabetes mellitus,immunosuppressive disorders)

  * Pregnant or lactating women
  * Heavy Smokers
  * Ongoing orthodontic treatment in the affected area
  * Use of medications affecting gingiva (e.g., phenytoin, cyclosporine, calcium channel blockers)
  * Poor oral hygiene at baseline
  * Active periodontal pockets >3 mm or clinical attachment loss
  * Allergy to local anesthetics or materials used in the procedure
  * History of alcohol or drug abuse
  * Psychological conditions that may interfere with compliance

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
gingival pigmentation intensity | Baseline, 1 Week, 1 month and at 3 months
  Dummett Oral Pigmentation Index (DOPI). This is an ordinal index that categorizes pigmentation on a 4-point scale: 0 = no pigmentation, 1 = mild, 2 = moderate, and 3 = heavy pigmentation.

SECONDARY OUTCOMES:
Patient Satisfaction | At Baseline, and at 3 months.
  Evaluated using a Visual Analog Score based questionnaire reflecting the Oral Health Related Quality of Life (OHRQoL), adapted from OHIP-1 to OHIP-14, measuring satisfaction with esthetic and functional outcomes following treatment. containing seven first-order factors (dimensions: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap) This instrument has a 5-point Likert-type response scale (0: never, 1: hardly ever, 2: occasionally, 3: fairly often, 4: very often).
Operating Time | Perioperative. From the start of the depigmentation procedure until the end of hemostasis and final inspection.
  Measured in minutes using a digital stopwatch from the start of the depigmentation procedure until the end of hemostasis and final inspection.
Pain Perception | Day 1, Day 3, 1 week, Day 10
  Assessed using a Visual Analog Scale (VAS), where participants will rate their pain perception on a continuous scale from 0 (no pain) to 10 (worst imaginable pain).
Extent of Pigmentation | Baseline, 1 Week, 1 month and at 3 months
  Assessed using the Takashi Index, a 3-grade ordinal scale scoring the extent of pigmentation as follows:0 = no pigmentation, 1 = isolated spots, and 2 = continuous ribbon. This will be recorded at each time point to assess reduction in pigmentation area.
Wound Healing | 1 week, 3 months
  Evaluated using the Healing Index of Landry, Turnbull, and Howley (1988), a 5-point scale ranging from 1 (very poor) to 5 (excellent), based on clinical observations of tissue color, bleeding, granulation, and epithelialization.
Recurrence Rate | 1 week, 1 month, and 3 months.
  Measured using the Melanin Pigmentation Index (MPI) at 1 week, 1 month, and 3 months postoperatively, scored as 0 = no pigmentation and 1 = presence of pigmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Darhous, Professor, Study Director — Cairo Univeristy; Maie Esmaiel, Lecturer, Study Chair — Cairo University; Raghad Hamadh, Bachelor, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt